CLINICAL TRIAL: NCT00676182
Title: Telerehabilitation for OIF/OEF Returnees With Combat-Related Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDR 08-267; a14714 (Other: United States: Federal Government)
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury; Post-traumatic Stress Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Telerehabilitation: telerehabilitation
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Rehabilitation via computer assisted internet capabilities

SUMMARY:
The scientific objective of this program is to meet the rehabilitation needs of combat wounded Veterans with mild to moderate Traumatic Brain Injury (TBI) via telerehabilitation and determine the effect of this modality of care on patients' physical health and outcomes including function and community participation. The investigators will also evaluate the benefits and limitations of rehabilitation using telehealth from the Veteran and caregiver perspectives and evaluate the impact of rehabilitation via telehealth on Veterans Administration (VA) healthcare facility use.

DETAILED DESCRIPTION:
Rational: TBI can cause life-long impairments in physical, cognitive, behavioral and social function that are usually more disabling than the residual physical deficits. Recovery can continue many years after initial trauma. Little is known about optimal methodologies to treat the vast and complicated secondary manifestations of combat related TBI. Applicability: The goal of this rehabilitation program is eventually to optimally define telerehabilitation services for all Veterans with polytrauma, including accurate and efficient screening instruments, educational material for patients and families, family support, and family counseling to enhance care coordination and to maximize functional outcomes and quality of life.

Patient population: The program will help wounded Veterans with a diagnosis of TBI from combat operations in Iraq and Afghanistan. Many Veterans reside in rural and underserved areas. Although access to health care for rural patients remains a critical challenge, telerehabilitation may represent a viable means for the delivery of therapeutic services to such patients, particularly those served by the VA. The program has implications for civilian populations as well including those injured in automobile or industrial accidents and similar in illness to the cohort of Veterans the investigators intend to follow.

Clinical applications, benefits and risks: The goals of the rehabilitation project will be to enhance the wounded Veteran's capacity to process and interpret information and to improve his ability to function in all aspects of family and community life. It will involve a combination of restorative training which focuses on improving a specific cognitive function and compensatory training which educates Veterans on adapting to the presence of a cognitive deficit that may or may not be curable using singular one to one interventions as well as integrated interdisciplinary approaches to target multiple conditions. The investigators see no risks involved in this clinical intervention.

Projected time to achieve a consumer-related outcome: The results of the telerehabilitation project should immediately be available for dissemination throughout the VA. The VA has already committed itself to a nationwide rollout of similar telerehabilitation projects for wounded Veterans. Hence, the findings should have immediate application in VA care for returnees from combat.

The investigators recently added MyHealtheVet to the TeleRehab I care coordination for existing TeleRehab I subjects. MyHealtheVet is the VA's Personal Health Record and offers Veterans an additional way for Veterans to partner with the health care team in making informed decisions. MyHealtheVet is an existing, innovative program available to Veterans throughout the VA. (see https://www.myhealth.va.gov/index.html for additional information) Most of the remaining TeleRehabilitation Veterans are already enrolled in the MyHealtheVet program. Besides giving patients access to their health records and online prescription ordering, there is a secure messaging system with VA providers, who can save the secure message into the patient's electronic medical record (CPRS) with a single click.

A total of 75 of the 85 IRB-approved subjects were initially enrolled. The investigators wanted to enroll up to 10 new subjects, and the existing TeleRehab I subjects were all be asked to sign a revised ICF that adds MyHealtheVet to the study, and makes other changes to the ICF required by Tampa VA R&D. If the subjects consent they will be required to register and be authenticated to use MyHealtheVet in order to participate or continue to participate in the study. An additional 6 subjects were enrolled for a total of 81 subjects on whom demographic data was collected. Sufficient data was collected on 75 subject for analyses of their responses to surveys.

MyHealtheVet enrollment and secure messaging authentication is required to continue in the study, and changes to the protocol will reflect this additional eligibility criterion. All other methods of communication with subjects and existing surveys will continue. Eventually MyHealtheVet will replace the LAMP for secure communications with the Care Coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Veterans or active duty military personnel discharged from the James A. Haley Veterans' Hospital in Tampa, FL or in rehabilitation there
* ages 18 and older
* have sustained a TBI as evidenced by primary or secondary diagnosis on initial admission, with or without comorbid Post-traumatic Stress Disorder (PTSD)
* enrolled and receiving medical services through the Tampa VA and medically stable as clinically determined by the patient's physician.

In order to add MyHealtheVet to the study as a method of care coordination, MyHealtheVet enrollment and secure messaging authentication is required to continue in the study. All other methods of communication with subjects and existing surveys will continue. Eventually MyHealtheVet will replace the LAMP for secure communications with the Care Coordinator.

Exclusion Criteria:

* Telerehab services will be offered only to those patients with low ADLs who require additional care and who stand to benefit from the care coordination program.
* The investigators will also exclude those who are severely injured or institutionalized. This includes patients with a severe psychopathology.
* Refusal to enroll in MyHealtheVet with Secure Messaging will eventually lead to subjects being dropped from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Convenience sample of OIF/OEF Veterans discharged from the James A. Haley Veterans' Hospital in Tampa, FL with a diagnosis of mild/moderate TBI with or without comorbid PTSD.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2008-07; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kris Siddharthan, PhD MS, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chapman PL, Elnitsky CA, Thurman R, Spehar AM, Siddharthan K. Exploring combat-related loss and behavioral health among OIF/OIF Veterans with chronic PTSD. Traumatology. 2013 Jun 1; 19(2):154-157.
- [Result] Siddharthan K. The effect of post traumatic stress disorders on rehabilitation among combat-wounded veterans. Stud Health Technol Inform. 2012;182:114-24. PMID 23138086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 participants were enrolled, but some did not participate or dropped out, leaving 75 participants who participated enough to collect data.
Groups:
- Telerehabilitation: telerehabilitation
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities
Period: Overall Study
Arm/Group | Telerehabilitation
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Telerehabilitation TBI: Telerehabilitation TBI
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities for veterans with TBI
- Telerehabilitation TBI/PTSD: Telerehabilitation TBI/PTSD
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities for veterans with TBI and comorbid PTSD
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation TBI | Telerehabilitation TBI/PTSD | Total
Number analyzed (Participants) | 61 | 14 | 75
Age, Customized [Number; unit: participants]
  18-29 years | 36 | 3 | 39
  30-39 years | 15 | 3 | 18
  40-49 years | 7 | 7 | 14
  50+ years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 58 | 14 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39 | 8 | 47
  Black | 4 | 0 | 4
  Hispanic | 15 | 4 | 19
  Native Hawaiian | 1 | 1 | 2
  Unanswered | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 61 | 14 | 75
Service Connected Disability Rating [Number; unit: participants] — Percent of service-connected disability
  participants
    0% | 17 | 5 | 22
    10-30% | 10 | 0 | 10
    40-60% | 14 | 3 | 17
    70-80% | 9 | 3 | 12
    80-100% | 11 | 3 | 14
Annual Income [Number; unit: participants]
  $0-9999 | 18 | 3 | 21
  $10,000-29,999 | 25 | 6 | 31
  $30,000-49,999 | 13 | 4 | 17
  $50,000-79,999 | 2 | 1 | 3
  $80,000+ | 3 | 0 | 3
Marital status [Number; unit: participants]
  Married | 32 | 7 | 39
  Divorced | 5 | 1 | 6
  Never Married | 20 | 6 | 26
  Single | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Functional Independence MeasureTM (FIM)/Functional Assessment Measure (FAM) (Total Score)
Description: Range: 30 - 210 FIMFAM Total Score: Higher value indicates higher function.
Time Frame: Baseline, 6 months, 12 months
Population: Only participants with data at the specified time points are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telerehabilitation: Telerehabilitation
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities for all subjects
Arm/Group | Telerehabilitation
Number analyzed (Participants) | 65
units on a scale
  Baseline (N=65) | 175.7 (33.7)
  6 Months (N=51) | 176.3 (29.8)
  12 Months (N=47) | 177.6 (26.7)

2. Primary Outcome: Craig Handicap Assessment and Reporting Technique (CHART)
Description: Ranges for Subscales: 0 - 100 Physical Independence: 4 -100 Cognitive Independence: 0 -100 Mobility: 0 -100 Occupation: 0 -100 Social Integration: 0 -100 Economic Self Sufficiency: 0-100
  Directionality: for each subscale, higher score means more independence; lower score means needs more assistance.
Time Frame: Baseline, 6 Months, 12 Months
Population: Only participants with data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telerehabilitation Baseline; Telerehabilitation 6 Months; Telerehabilitation 12 Months: telerehabilitation
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities
Arm/Group | Telerehabilitation Baseline | Telerehabilitation 6 Months | Telerehabilitation 12 Months
Number analyzed (Participants) | 66 | 51 | 47
units on a scale
  Physical Independence | 85.4 (34.5) | 87.3 (28.5) | 70.5 (117.1)
  Cognitive Independence | 66.8 (28.5) | 58.1 (29.4) | 63.4 (30.2)
  Mobility | 79.6 (24.1) | 78.9 (23.4) | 79.2 (25)
  Occupation | 69.8 (36.9) | 71 (36.6) | 73.1 (38.8)
  Social Integration | 84.4 (22.2) | 76.1 (25.9) | 82.5 (21.4)
  Economic Self Sufficiency | 81 (24.2) | 79.7 (27.2) | 77.4 (26.5)

3. Primary Outcome: Patient Competency Rating Scale (PCRS) (Total Score)
Description: Range for total score: 30 - 150 Directionality for total score: higher score means higher competency (can do things with greater ease)
Time Frame: Baseline, 6 Months, 12 Months
Population: Only participants with data at the specified time were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation
Number analyzed (Participants) | 66
units on a scale
  Baseline (N=66) | 91 (16.2)
  6 Months (N=51) | 90.9 (20.6)
  12 Months (N=45) | 94.4 (21.1)

4. Primary Outcome: PTSD Checklist Military Form (PCL-M) (Total Score)
Description: Range for total score: 17- 85 Directionality for total score: Higher score means experiencing more PTSD-related problems.
Time Frame: Baseline, 6 Months, 12 Months
Population: Veterans with TBI with comorbid PTSD who were analyzed at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telerehabilitation TBI/PTSD: telerehabilitation
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities for TBI/PTSD
Arm/Group | Telerehabilitation TBI/PTSD
Number analyzed (Participants) | 14
units on a scale
  Baseline (N=14) | 63.6 (10.6)
  6 Months (N=11) | 64.1 (14)
  12 Months (N=10) | 59.4 (12.4)

5. Primary Outcome: Modified PTSD Symptom Scale: Self-Report - Frequency (Total Score)
Description: Range for Total Score: 0-68 Directionality: Higher score means more PTSD-related symptoms.
Time Frame: Baseline, 6 Months, 12 Months
Population: Veterans with TBI and comorbid PTSD with data at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telerehabilitation TBI/PTSD: telerehabilitation
  Telerehabilitation: Rehabilitation via computer assisted internet capabilities for veterans with TBI/PTSD
Arm/Group | Telerehabilitation TBI/PTSD
Number analyzed (Participants) | 14
units on a scale
  Baseline (N=14) | 54.2 (8.5)
  6 Months (N=11) | 53.3 (11.5)
  12 Months (N=10) | 49.1 (14.4)

6. Primary Outcome: Modified PTSD Symptom Scale: Self-Report - Severity
Description: Range for Total Score: 0 - 68 Directionality: Higher score means more PTSD-related symptoms.
Time Frame: Baseline, 6 Months, 12 Months
Population: Only veterans with TBI and comorbid PTSD with data at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation TBI/PTSD
Number analyzed (Participants) | 14
units on a scale
  Baseline (N=14) | 64.1 (14.3)
  6 Months (N=11) | 62.7 (17.8)
  12 Months (N=10) | 55.3 (20.6)

7. Primary Outcome: Alcohol Use Disorders Identification Test (AUDIT) (Total Score)
Description: Range for Total Score: 0-40 Directionality: Higher score means more alcohol use.
Time Frame: Baseline, 6 Months, 12 Months
Population: Only veterans with TBI and comorbid PTSD with data at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation TBI/PTSD
Number analyzed (Participants) | 14
units on a scale
  Baseline (N=14) | 5.1 (7.2)
  6 Months (N=11) | 4.8 (5.6)
  12 Months (N=10) | 6 (5.6)

8. Primary Outcome: Beck Depression Inventory Score (Total Score)
Description: Range for Total Score: 0-63 Directionality: Higher score means more depression-related symptoms.
Time Frame: Baseline, 6 Months, 12 Months
Population: Only veterans with TBI and comorbid PTSD with data at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation TBI/PTSD
Number analyzed (Participants) | 14
units on a scale
  Baseline (N=14) | 33.1 (13.6)
  6 Months (N=11) | 33.7 (13.7)
  12 Months (N=10) | 30.6 (11.8)

ADVERSE EVENTS:
Arm/Group | Telerehabilitation
Serious Adverse Events (participants affected / at risk) | 4/75
Other Adverse Events (participants affected / at risk) | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation (N=75)
Death (General disorders) | 1 (1)
Hospitalization due to suicidal ideation (General disorders) | 1 (1)
Hospitalization (General disorders) | 1 (1) — event leading to hospitalization unknown
Hospitalization (General disorders) | 1 (1) — event unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No